CLINICAL TRIAL: NCT06544265
Title: A Phase 1 Study of SynKIR-310, Autologous T Cells Transduced With CD19 KIR-CAR, in Participants With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: SynKIR-310 for Relapsed/Refractory B-NHL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Verismo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CELESTIAL-301
Record Dates: First submitted 2024-07-11; First posted 2024-08-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: B Cell Lymphoma; NHL, Adult; Mantle Cell Lymphoma; Relapsed Non-Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; Aggressive B-Cell Non-Hodgkin Lymphoma; Indolent B-Cell Non-Hodgkin Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; DLBCL - Diffuse Large B Cell Lymphoma; HGBL With MYC and BCL2 and/or BCL6 Rearrangements; High-grade B-cell Lymphoma; Diffuse Large B Cell Lymphoma; Large B-cell Lymphoma; T-Cell/Histiocyte Rich Lymphoma; Non-hodgkin Lymphoma,B Cell; Primary Mediastinal Large B-cell Lymphoma (PMBCL); Epstein-Barr Virus Positive DLBCL, Nos; Follicular Lymphoma Grade 3B; DLBCL (Diffuse Large B-Cell Lymphoma) Associated With Chronic Inflammation; High Grade B-Cell Lymphoma, Not Otherwise Specified; Follicular Lymphoma Grade 3; Marginal Zone Splenic Lymphoma; DLBCL
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Large B-Cell, Diffuse; Pyloric Stenosis, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SynKIR-310 (Experimental): Single dose IV administration of SynKIR-310
  Interventions: Biological: SynKIR-310

INTERVENTIONS:
Biological: SynKIR-310 — Autologous T Cells transduced with CD19 KIR-CAR

SUMMARY:
This first-in-human (FIH) trial is designed to assess the safety, feasibility and preliminary efficacy of a single intravenous (IV) dose of SynKIR-310 administered to participants with relapsed/refractory B-NHL.

DETAILED DESCRIPTION:
This is a Phase 1, FIH, multicenter, open-label study of a single infusion of SynKIR-310 in participants with relapsed/refractory B-NHL.

Up to 18 participants, regardless of subtypes of B-NHL, who meet the eligibility criteria, will be treated in the study.

2 cohorts of 3 to 6 participants per cohort will be assessed to determine the safety and feasibility of treatment with SynKIR-310. Doses will be escalated across 2 cohorts to determine a Recommended Phase 2 Dose (RP2D).

Once the RP2D has been determined, a dose expansion group will enroll additional participants regardless of subtypes of B-NHL at the RP2D to further characterize the safety, feasibility and preliminary efficacy of SynKIR-310 in treating B-NHL.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years of age and older.
* Histologically confirmed diagnosis of B-NHL before enrollment.
* Must have received prior CAR T or were unwilling/unable to receive prior CAR T.
* Must have refractory or relapsed disease after receiving 2 prior lines of therapies.
* If relapsed/refractory post-auto-SCT, then must have undergone auto-SCT at least 6 months prior to enrollment.
* If relapsed/refractory disease after allogeneic stem cell transplant (allo SCT) then must have undergone allo-SCT at least 6 months prior to enrollment and without evidence of graft versus host disease.
* Measurable disease at time of enrollment: At least one measurable lesion per Lugano Response Criteria (Cheson et al., 2014).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1

Exclusion Criteria:

* Previously treated with any investigational agent within 30 days prior to screening.
* Adequately treated non-melanoma skin cancer such as basal cell or squamous cell carcinoma
* Carcinoma-in-situ (e.g., cervix, bladder, breast) treated curatively and without evidence of recurrence for at least 3 years prior to enrollment.
* Any other malignancy which has been completely treated and remains in complete remission for ≥ 5 years prior to enrollment. Completely treated prostate cancer with prostate-specific antigen (PSA) level < 1.0 may also be permitted.
* Known immunodeficiency disease.
* History or presence of active or clinically relevant primary central nervous system (CNS) disorder, such as seizure, encephalopathy, cerebrovascular ischemia/hemorrhage, cerebellar disease, or any autoimmune disease with CNS involvement. For primary CNS disorders that have recovered or are in remission, participants without recurrence within 2 years of planned study enrollment may be included.
* Uncontrolled hypertension, history of myocarditis or congestive heart failure, unstable angina, serious uncontrolled cardiac arrhythmia, or myocardial infarction within 6 months prior to study entry.
* Any active uncontrolled systemic fungal, bacterial or viral infection.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of SynKIR310 | Up to 24 months
  The incidence, frequency, and severity of adverse events (AEs), including serious adverse events (SAEs), treatment-emergent adverse events (TEAEs), and dose-limiting toxicities (DLTs).
Recommended Phase 2 Dose (RP2D) | Up to 24 months
  All available data from dose escalation cohorts will be evaluated to determine RP2D

SECONDARY OUTCOMES:
Feasibility of SynKIR-310 | Up to 24 months
  Number of enrolled patients who receive SynKIR-310.
Preliminary efficacy : Objective response rate (ORR) | Up to 24 months
  Percentage of patients with a complete or partial response determined by Investigator
Preliminary efficacy: Complete response rate (CR) | Up to 24 months
  Percentage of patients with a Complete Response determined by Investigator
Preliminary efficacy: Duration of response (DOR) | Up to 24 months
  Time from the date of the first occurrence of complete response or partial response to the date of progression, relapse, or death from any cause, determined by Investigator
PD profile of SynKIR-310 | Up to 24 months
  To evaluate concentration of cytokines in serum over time following SynKIR-310 infusion
PK profile of SynKIR-310 | Up to 24 months
  To evaluate the patients who show CAR T persistence in blood (measured in the blood by quantitative polymerase chain reaction (PCR)) at multiple study time points following SynKIR-310 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Johnson, PhD, Study Chair — Verismo Therapeutics
Locations (5):
- United States (5):
  - Colorado Blood Cancer Institute, part of Sarah Cannon Cancer Institute, Denver, Colorado
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - The University of Kansas Cancer Center, Fairway, Kansas
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No